CLINICAL TRIAL: NCT05036707
Title: Investigating the Human Immune Response to Ixodes Scapularis Tick Bites
Brief Title: Human Immune Response to Ixodes Scapularis Tick Bites
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000331; 000331-I
Record Dates: First submitted 2021-09-04; First posted 2021-09-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05-16

CONDITIONS: Tick-borne Diseases; Tick Resistance; Lyme Disease
Keywords: Tick Immunity; Tick-borne diseases; Vaccines; Lyme Disease
MeSH Terms: conditions — Tick-Borne Diseases; Lyme Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 1 (Active Comparator): Healthy Volunteer
  Interventions: Device: Xenodiagnosis Ticks; Procedure: skin biopsy; Procedure: blood draw

INTERVENTIONS:
Device: Xenodiagnosis Ticks — Larval ticks will be obtained from Dr. Sam Telford from a laboratory maintained tick colony at Tufts Veterinary School. These ticks are hatched from eggs laid by ticks that have fed only on specific pathogen free laboratory animals that were purchased from established vendors.
Procedure: skin biopsy — 2-3 mm skin punch biopsies will be performed.
Procedure: blood draw — Peripheral blood draws will be performed.

SUMMARY:
Background:

Each year, the number of cases of tick-borne diseases increases. The deer tick (Ixodes scapularis) is the vector of at least 7 pathogens that cause human diseases, including Lyme disease. Researchers want to learn more to help them develop vaccines against ticks in the future.

Objective:

To learn how people s bodies, particularly the skin, respond to tick bites.

Eligibility:

Healthy adults aged 18 years and older who have no known history of a tick-borne disease or tick bite exposure.

Design:

Participants will be screened with a medical history, physical exam, and blood tests.

Participants will have 2 skin punch biopsies of healthy skin. For this, a sharp instrument will be used to remove a round plug of skin about the size of a pencil eraser. Participants will then have 10 clean laboratory-bred ticks placed at 2 different sites on their skin (20 ticks total). The ticks will be removed from the first site 1 day after placement and from the second site 2-4 days after placement. Participants will complete symptom diary cards. They will answer questions about itching at the tick feeding sites. They will give blood samples. Photos will be taken of the tick feeding sites. Skin punch biopsies will be collected at the sites of the tick bites.

Participants will repeat the tick feeding procedures 2 times, each 2-8 weeks apart. For the 2nd and 3rd procedures, 10 clean laboratory-bred ticks will be placed at 1 site. The ticks will be removed 2-3 days after tick placement. They will have telephone follow-up visits after each procedure.

After the final tick removal, participants will have follow-up visits in 4-6 weeks and again in 3 months. They will give blood samples and discuss how they are feeling.

Participation will last about 5-7 months.

DETAILED DESCRIPTION:
Study Description:

This study aims to develop a model for acquired tick resistance in humans, characterize the acquisition of tick-associated skin immunity, and monitor the innate and adaptive immune response of Ixodes scapularis tick bites. The study will be a prospective, non-randomized, single-center study performed at the National Institutes of Health (NIH) Clinical Center. It will be performed under Investigational Device Exemption (IDE) G210153, and will be monitored as per National Institute of Allergy and Infectious Diseases (NIAID) and NIH regulations. Participants (35 adult healthy volunteers) will undergo up to 3 tick feeding placements, 2 to 8 weeks

apart. One to two punch skin biopsies (2-3 mm) from the tick bite sites will be collected at 1 day (early) and 2-4 days (late) after the first tick placement procedure. Skin biopsies of an unaffected site will be performed as a control. One to two punch skin biopsies (2-3 mm) from the tick bite sites will be collected at day 2-3 after the 2nd and 3rd tick placement procedures. Additionally, blood will be collected to evaluate systemic immune response to tick salivary proteins. Ticks will also be collected at each timepoint and gene expression will be analyzed to determine the effect of the human skin response on ticks.

Changes in resistance to tick bites can be evaluated by:

* Local reaction to the tick bite

  * pruritus
  * site reactions
  * Blood flow index as measured by laser speckle contrast imaging
* Number of fed ticks

Changes in the immune response and cellular recruitment in the skin can be evaluated using:

Differential expression of immune transcripts and other skin associated transcripts using RNAseq or other high-throughput profiling of cells

Conventional histology and immunohistochemistry

Digital Spatial Profiling to determine cell type and other immune markers using a high-plex platform

Changes in the systemic immune response will be evaluated by:

Measurement of antibodies against tick salivary proteins will be assessed by enzyme-linked immunosorbent assay (ELISA) and

western blot

Novel state-of-the-art high resolution technologies to deeply characterize the immune response to tick bites over time, both phenotypically and functionally.

Changes in tick transcriptomic profile will be assessed by:

RNAseq: Ribonucleic acid (RNA) will be isolated from tick after they have been removed from subjects and unexposed ticks.

Differential expression profile will be performed and validated by NanoString

Objectives:

Primary Objectives:

1. Develop a model of acquired tick resistance in humans
2. Continue to assess the safety of tick feeding using laboratory-reared Ixodes scapularis larva in humans

Exploratory Objectives:

1. Comparison of the early and late immune response in the skin site of the bite of Ixodes scapularis after a single tick exposure.
2. Determine the effects of repeated tick feeding on the immune response at the tick bite site in human skin and development of tick resistance.
3. Analyze the evolution of the systemic immune response to tick bite in participants after multiple tick exposures and validate development of reliable biomarkers of tick exposure.
4. Analyze gene expression of Ixodes scapularis larvae feeding on humans and determine the effects of immune response of subjects

repeatedly bitten on larvae gene expression.

Endpoints:

Primary Endpoints:

1. Pruritus at the site of tick attachment in the first 24 hours of tick placement over the three placements as measured by a positive slope

   over the three placements of the numerical rating score. The slope of other pruritus scores at 24 hours and at Day 2-4, and the number of attached ticks collected from participants over the three placements will also be measured.
2. Monitor safety adverse events (AEs) using reporting tools and Sponsor safety monitors.

Exploratory Endpoints:

1. Compare the results from the skin biopsies acquired with the first tick placement. Our hypothesis is that there will be differential phenotypic, transcriptomic, and immunohistochemical differences between:

   * Exposed (bitten skin at day 1) and unexposed (unbitten skin)
   * Exposed (bitten skin at day 2-4) and unexposed (unbitten skin)
   * Exposed (bitten skin at day 1) and exposed (bitten skin at day 2-4)

   Measurement of changes will be assessed by:
   * Differential expression of immune transcripts and other skin associated transcripts using RNAseq
   * Conventional histology and immunohistochemistry
   * Digital Spatial Profiling to determine cell type and other immune markers using a high-plex platform
2. Compare the changes in the local immune response and cellular recruitment between the 1st, 2nd and the 3rd tick exposures and correlate with measures of itching, blood flow index and number of attached ticks and the feeding status.

   We postulate that differences between the timepoints will become more marked with multiple exposures. We hypothesize that there will be differential phenotypic and transcriptomic differences between:

   Exposed (bitten skin at day 2-3, exposure 2) and exposed (bitten skin at day 2-3, exposure 3)

   Correlate these changes with measures of resistance to tick feeding (itching, number and level of feeding of attached ticks, blood flow index).
3. Compare the development of antibody responses against Ixodes scapularis salivary protein antigens between the 1st, 2nd, and the 3rd tick exposures and correlate antibodies against tick salivary proteins with measures of resistance (itching, erythema, blood flow index, number of fed ticks).

   Explore the development of the host response in blood using high resolution technologies such as immunophenotyping, proteomics and

   transcriptomics and compare the responses between the 1st, 2nd, and the 3rd tick exposures.
4. Using RNAseq technology, measure changes in gene expression of ticks fed at early timepoint (1 day) vs late timepoint (2-4 days) vs unfed ticks and of ticks fed at 1st, 2nd, and 3rd placements. Correlation of pruritus and changes in tick gene expression.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Age 18 years or older.
3. In good general health as evidenced by medical history.
4. No history of TBD.
5. No known tick bite.
6. Serum IgE level within Clinical Center Department of Laboratory Medicine normal range.

   https://ccinternal2.cc.nih.gov/LTGRA/UL/public_labtest_detail.aspx?next_flg=Y&test_id=4731&id_order=53
7. Serum tryptase level within Clinical Center Department of Laboratory Medicine normal range.

   https://ccinternal2.cc.nih.gov/LTGRA/UL/public_labtest_detail.aspx?next_flg=Y&test_id=1157&id_order=1
8. For participants of child-bearing potential: use of effective contraception for at least 1 month prior to tick placement, and agreement to use such a method during study participation and for an additional 3 months after the removal of the last ticks. Types of contraception include abstinence, surgical methods (sterilization, implants, intrauterine device, partner with vasectomy), hormonal methods (birth control pill, patch, ring, injection), or barrier methods (diaphragm plus spermicide, male condom plus spermicide)
9. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
10. Agree to not participate in other clinical studies requiring investigational interventions for the duration of the study.
11. Minimum hemoglobin of 13.0 g/dL for males and 12 g/dL for females

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of forming large thick scars (keloids) after skin injuries.
2. History of excessive bleeding after cuts or procedures.
3. History of taking anticoagulants in the past 28 days.
4. History of allergic reaction to lidocaine.
5. History of allergic reaction to tape, adhesive bandages, or dressings.
6. Inability to maintain the dressing for any reason.
7. Pregnancy or lactation.
8. Treatment with another investigational drug or other intervention within the past 30 days.
9. Oral or intravenous (IV) steroids in the 2 weeks prior to each tick placement procedure (topical, nasal, inhaled, intra-articular, and replacement doses of steroids are not exclusions).
10. History of reactions to mammalian meat, IgE- mediated food allergies, urticaria or anaphylaxis. Mild pollen-food allergy syndrome is not an exclusion.
11. History of systemic allergic reaction to venom (bee, wasps and other Hymenoptera stings).
12. History of clinically significant drug allergies.
13. History of moderate to severe atopy asthma, atopic dermatitis, allergic rhinitis.
14. Active severe skin disease, uncontrolled diabetes, cancer other than non-melanoma skin cancers, autoimmune disease requiring immunosuppressive therapy, or history of human immunodeficiency virus (HIV), chronic viral hepatitis, or syphilis.
15. Refusal to allow storage of samples and data for future usage..
16. Any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in and completing the study.

Exclusion of Select Populations:

Children:

Children are excluded from this protocol as there is no direct benefit to the participants, the risk from the skin biopsies is small but above minimal, the procedure is invasive and can be stressful for children, and there is concern over their ability to maintain the LeFlap dressing.

Pregnant and breastfeeding women:

Pregnant and breastfeeding women are excluded from trial participation as there is no direct benefit to the participants.

Adults who lack capacity to consent:

Adults lacking decision-making capacity to provide informed consent are excluded at screening as there is no direct benefit to the participants.

Enrolled participants who permanently lose the ability to consent during participation will be monitored for safety but will have no additional research procedures performed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Safety of the device. Use toxicity tables and safety monitoring as specified in the protocol. | continuous
  Ongoing assessment of safety.
Develop a model of acquired tick resistance in humans. Use validated pruritus scales, numerical rating system, verbal rating system, and visual analogue system. | end of study
  Clinical measures of tick immunity.

SECONDARY OUTCOMES:
Exploratory: Determine the effects of repeated tick feeding on immune response at tick bite site and the development of resistance. Use RNASeq,histology, immunohistochemistry, digital spatial profiling, clinical itch scales, site reactions, tick... | continuous
  Compare changes in early and late local immune response and cellular recruitment between the 1st and 3rd tick exposures.
Exploratory: Analyze gene expression of Ixodes scapularis after feeding on humans using RNASeq. | continuous
  Measure changes in gene expression of ticks fed at the various time points.
Exploratory: Compare early and late immune response in skin after Ixodes scapularis bite. Use RNASeq, histology, immunohistochemistry, digital spatial profiling to explore. | continuous
  Compare early and late immune response in the skin using skin biopsies collected at Day 1 and Day 4.
Exploratory: Analyze the evolution of the systemic immune response to tick bite by measuring antibodies response (ELISA and western blot) against Ixodes scapularis salivary protein antigens. | continous
  Compare the development of antibody responses against Ixodes scapularis salivary antigens between the 1st, 2nd, and 3rd tick feedings.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if the research results will reveal a need to disclose IPD, therefore it is undecided if we plan to make IPD available.

REFERENCES:
- [Background] Marques A, Telford SR 3rd, Turk SP, Chung E, Williams C, Dardick K, Krause PJ, Brandeburg C, Crowder CD, Carolan HE, Eshoo MW, Shaw PA, Hu LT. Xenodiagnosis to detect Borrelia burgdorferi infection: a first-in-human study. Clin Infect Dis. 2014 Apr;58(7):937-45. doi: 10.1093/cid/cit939. Epub 2014 Feb 11. PMID 24523212
- [Background] Ribeiro JM, Alarcon-Chaidez F, Francischetti IM, Mans BJ, Mather TN, Valenzuela JG, Wikel SK. An annotated catalog of salivary gland transcripts from Ixodes scapularis ticks. Insect Biochem Mol Biol. 2006 Feb;36(2):111-29. doi: 10.1016/j.ibmb.2005.11.005. Epub 2005 Dec 20. PMID 16431279
- [Background] Valenzuela JG. Exploring tick saliva: from biochemistry to 'sialomes' and functional genomics. Parasitology. 2004;129 Suppl:S83-94. doi: 10.1017/s0031182004005189. PMID 15938506
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000331-I.html